CLINICAL TRIAL: NCT03153345
Title: The Efficacy of Bedside Respiratory Muscle Training in Stroke Patients: A Randomized Controlled Trial
Brief Title: The Efficacy of Bedside Respiratory Muscle Training in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Joon Yoo, Principal Investigator, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KoreaUAnamHRehab
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Stroke; Rehabilitation; Breathing Exercise; Pneumonia; Respiration
MeSH Terms: conditions — Stroke; Pneumonia; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Experimental): The intervention group participated in a conventional stroke rehabilitation program, which consisted of joint range of motion exercises, muscle strengthening, gait training, fine motor exercises, and activity of daily living training. This program was performed for 30 minutes twice a day 5 days a week, over for at least 3 weeks. During the same period, the intervention group also took part in bedside respiratory muscle training twice a day for 7 days a week over a 3-week period.
  Interventions: Device: bedside respiratory muscle training; Behavioral: conventional stroke rehabilitation program
- Control group (Active Comparator): The control group participated only in a conventional stroke rehabilitation program, which consisted of joint range of motion exercises, muscle strengthening, gait training, fine motor exercises, and activity of daily living training. This program was performed for 30 minutes twice a day 5 days a week, over for at least 3 weeks.
  Interventions: Behavioral: conventional stroke rehabilitation program

INTERVENTIONS:
Device: bedside respiratory muscle training — The program consisted of three sessions: (1) 10 minutes of breath stacking exercise, followed by (2) 10 minutes of inspiratory muscle training using a flow-oriented incentive spirometer and (3) 10 minutes of expiratory muscle training using Acapella vibratory PEP device.
  Arms: Intervention group
Behavioral: conventional stroke rehabilitation program — The program consisted of joint range of motion exercises, muscle strengthening, gait training, fine motor exercises, and activity of daily living training.

SUMMARY:
Objectives: To investigate the efficacy of bedside respiratory muscle training on pulmonary function and stroke-related disabilities in stroke patients.

Design: Prospective randomized controlled trial

Setting: A single physical medicine and rehabilitation department at a university hospital

Participants: Stroke patients in a rehabilitation unit were recruited and randomly assigned to either the intervention group or the control group.

Intervention: Both groups participated in a conventional stroke rehabilitation program. During the study period, the intervention group received bedside respiratory muscle training twice a day for three weeks. The respiratory muscle training consisted of (1) a breath stacking exercise, (2) inspiratory muscle training and (3) expiratory muscle training. The participants were evaluated at baseline and again at the end of the study (3 weeks later).

Main Outcome Measures: The primary outcomes were measures of pulmonary function: functional vital capacity (FVC), forced expiratory volume in one second (FEV1) and peak flow.

Secondary outcomes were stroke-related disabilities assessed by the following: National Institutes of Health Stroke Scale, Modified Barthel Index, Berg Balance Scale, Fugl-Meyer Assessment, the Korean Mini-Mental State Examination, and the incidence of pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years of age,
2. first episode of stroke within three months,
3. moderate to severe stroke impairment, defined as a NIHSS score from 5-36, and
4. the ability to follow instructions and engage in the study program.

Exclusion Criteria:

1. a medical history of persistent cardiopulmonary disease,
2. other coexisting brain disorders, such as brain tumor,
3. poorly controlled hypertension, which was defined as a blood pressure higher than 180/100 mmHg during the preceding 24 hours,
4. severe facial palsy or other oropharyngeal structural abnormality,
5. severe oral apraxia, and (6) having a tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
functional vital capacity | 21 days
  functional vital capacity in percent (%)
Forced expiratory volume | 21 days
  Forced expiratory volume in one second in percent (%)
Peak flow | 21 days
  Peak flow in milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bom Pyun, M.D, Ph.D, Study Chair — Department of Physical Medicine and Rehabilitation, Korea University Anam Hospital, Korea University College of Medicine